CLINICAL TRIAL: NCT02163759
Title: Phase III, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy (Induction of Remission) and Safety of Etrolizumab Compared With Adalimumab and Placebo in Patients With Moderate to Severe Ulcerative Colitis Who Are Naive to TNF Inhibitors
Brief Title: A Study Comparing the Efficacy and Safety of Etrolizumab With Adalimumab and Placebo in Participants With Moderate to Severe Ulcerative Colitis (UC) in Participants Naive to Tumor Necrosis Factor (TNF) Inhibitors
Acronym: HIBISCUS I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA28948; 2013-004279-11 (EudraCT Number)
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Results first posted 2021-04-05 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab; etrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo matching to etrolizumab up to Week 12 and placebo matching to adalimumab up to Week 8.
  Interventions: Other: Adalimumab Placebo; Other: Etrolizumab Placebo
- Adalimumab (Active Comparator): Participants will receive adalimumab up to Week 8 and placebo matching to etrolizumab up to Week 12.
  Interventions: Drug: Adalimumab; Other: Etrolizumab Placebo
- Etrolizumab (Experimental): Participants will receive etrolizumab up to Week 12 and placebo matching to adalimumab up to Week 8.
  Interventions: Other: Adalimumab Placebo; Drug: Etrolizumab

INTERVENTIONS:
Drug: Adalimumab — Adalimumab 160 milligrams (mg) will be administered subcutaneously (SC) at Week 0; 80 mg SC at Week 2; 40 mg SC at Weeks 4, 6, and 8.
  Other Names: Humira
  Arms: Adalimumab
Other: Adalimumab Placebo — Placebo matching to adalimumab will be administered SC at Weeks 0, 2, 4, 6, and 8.
  Arms: Etrolizumab; Placebo
Drug: Etrolizumab — Etrolizumab 105 mg will be administered SC every 4 weeks (Q4W) up to Week 12 (at Weeks 0 [Day 1], 4, 8, and 12 [clinical remitters only]).
  Other Names: PRO145223; RO5490261; RG7413
  Arms: Etrolizumab
Other: Etrolizumab Placebo — Placebo matching to etrolizumab will be administered SC once every 4 weeks (Q4W) up to Week 12 (at Weeks 0 [Day 1], 4, 8, and 12 [clinical remitters only]).
  Arms: Adalimumab; Placebo

SUMMARY:
This Phase III, double-blind, placebo and active-comparator controlled, multicenter study will investigate the efficacy and safety of etrolizumab in induction of remission in participants with moderately to severely active ulcerative colitis (UC) who are naÏve to tumor necrosis factor (TNF) inhibitors and refractory to or intolerant of prior immunosuppressant and/or corticosteroid treatment. In addition to this study, a second Phase III trial with identical study design (GA28949; NCT02171429) was independently conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis (UC) established at least 3 months prior to randomization (Day 1)
* Moderately to severely active UC as determined by the MCS
* Naive to treatment with TNF inhibitor therapy
* An inadequate response, loss of response, or intolerance to prior corticosteroid and/or immunosuppressant treatment
* Background UC therapy may include oral 5-aminosalisylate (5-ASA), budesonide, oral corticosteroids, probiotics, azathioprine (AZA), 6-mercaptopurine (6MP), or methotrexate (MTX) if doses have been stable for:
* AZA, 6-MP, MTX: 8 weeks immediately prior to randomization
* 5-ASA: 4 weeks immediately prior to randomization
* Corticosteroids: 4 weeks immediately prior to randomization; if corticosteroids are being tapered, dose has to be stable for at least 2 weeks prior to randomization
* Use of highly effective contraception method as defined by the protocol
* Have received a colonoscopy within the past year or be willing to undergo a colonoscopy in lieu of a flexible sigmoidoscopy at screening

Exclusion Criteria:

Exclusion Criteria Related to Inflammatory Bowel Disease:

* Prior extensive colonic resection, subtotal or total colectomy, or planned surgery for UC
* Past or present ileostomy or colostomy
* Diagnosis of indeterminate colitis
* Suspicion of ischemic colitis, radiation colitis, or microscopic colitis
* Diagnosis of toxic megacolon within 12 months of initial screening visit
* Any diagnosis of Crohn's disease
* Past or present fistula or abdominal abscess
* A history or current evidence of colonic mucosal dysplasia
* Patients with any stricture (stenosis) of the colon
* Patients with history or evidence of adenomatous colonic polyps that have not been removed

Exclusion Criteria Related to Prior or Concomitant Therapy:

* Prior treatment with TNF-alpha antagonists
* Any prior treatment with etrolizumab or other anti-integrin agents
* Any prior treatment with rituximab
* Any treatment with tofacitinib during screening
* Any prior treatment with anti-adhesion molecules
* Use of intravenous (IV) steroids within 30 days prior to screening with the exception of a single administration of IV steroid
* Use of agents that deplete B or T cells
* Use of anakinra, abatacept, cyclosporine, sirolimus, or mycophenolate mofetil (MMF) within 4 weeks prior to randomization
* Chronic nonsteroidal anti-inflammatory drug (NSAID) use
* Patients who are currently using anticoagulants including, but not limited to, warfarin, heparin, enoxaparin, dabigatran, apixaban, rivaroxaban
* Patients who have received treatment with corticosteroid enemas/suppositories and/or topical (rectal) 5-ASA preparations within 2 weeks prior to randomization
* Apheresis (i.e., Adacolumn apheresis) within 2 weeks prior to randomization
* Received any investigational treatment including investigational vaccines within 5 half lives of the investigational product or 28 days after the last dose, whichever is greater, prior to randomization
* History of moderate or severe allergic or anaphylactic/anaphylactoid reactions to chimeric, human, or humanized antibodies, fusion proteins, or murine proteins or hypersensitivity to etrolizumab (active drug substance) or any of the excipients (L histidine, L-arginine, succinic acid, polysorbate 20)
* Patients administered tube feeding, defined formula diets, or parenteral alimentation/nutrition who have not discontinued these treatments within 3 weeks prior to randomization

Exclusion Criteria Related to General Safety:

* Pregnant or lactating
* Lack of peripheral venous access
* Hospitalization (other than for elective reasons) during the screening period
* Significant uncontrolled comorbidity, such as cardiac (e.g., moderate to severe heart failure New York Heart Association Class III/IV), pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders
* Neurological conditions or diseases that may interfere with monitoring for PML
* History of demyelinating disease
* Clinically significant abnormalities on screening neurologic examination (PML Objective Checklist)
* Clinically significant abnormalities on the screening PML Subjective Checklist
* History of alcohol, drug, or chemical abuse less than 6 months prior to screening
* Conditions other than UC that could require treatment with >10 mg/day of prednisone (or equivalent) during the course of the study
* History of cancer, including hematologic malignancy, solid tumors, and carcinoma in situ, within 5 years before screening

Exclusion Criteria Related to Infection Risk

* Congenital or acquired immune deficiency
* Patients must undergo screening for HIV and test positive for preliminary and confirmatory tests
* Positive hepatitis C virus (HCV) antibody test result
* Positive hepatitis B virus (HBV) antibody test result
* Evidence of or treatment for Clostridium difficile (as assessed by C. difficile toxin testing) within 60 days prior to randomization or other intestinal pathogens (as assessed by stool culture and ova and parasite evaluation) within 30 days prior to randomization
* Evidence of or treatment for clinically significant cytomegalovirus (CMV) colitis (based on the investigator's judgment) within 60 days prior to randomization
* History of active or latent TB
* History of recurrent opportunistic infections and/or history of severe disseminated viral infections
* Any serious opportunistic infection within the last 6 months prior to screening
* Any current or recent signs or symptoms (within 4 weeks before screening and during screening) of infection
* Any major episode of infection requiring treatment with IV antibiotics within 8 weeks prior to screening or oral antibiotics within 4 weeks prior to screening
* Received a live attenuated vaccine within 4 weeks prior to randomization
* History of organ transplant

Exclusion Criteria Related to Laboratory Abnormalities (at Screening)

* Serum creatinine >2 x upper limit of normal (ULN)
* ALT or AST >3 x ULN or alkaline phosphatase >3 x ULN or total bilirubin >2.5 x ULN
* Platelet count <100,000/uL
* Hemoglobin <8 g/dL
* Absolute neutrophil count <1500/uL
* Absolute lymphocyte count <500/uL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (88):
- United States (9):
  - Rocky Mountain Gastroenterology Associates, P.L.L.C.; Gastroenterology, Lakewood, Colorado
  - Center for Advanced Gastroenterology, Maitland, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Center for Digestive Health, Troy, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Wellness Clinical Research Center, San Antonio, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
- Instituto Medico DAMIC, Córdoba, Argentina
- Australia (6):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Brazil (6):
  - CCBR - Brasilia, Brasília, Federal District
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda, Goiânia, Goiás
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Hospital Universitario Clementino Fraga Filho - UFRJ, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
- Bulgaria (3):
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - UMHAT Tsaritsa Yoanna - ISUL, EAD, Sofia
  - MC Medica Plus, Veliko Tarnovo
- Estonia (5):
  - OÜ Innomedica, Tallinn
  - East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- France (2):
  - Hôpital Beaujon, Clichy
  - CHU Nice - Hopital de l'Archet 2, Nice
- University of Hong Kong, Hong Kong, Hong Kong
- Mexico (3):
  - Centro Integral en Reumatología S.A. de C.V. (CIRSA), Guadalajara, Jalisco
  - Accelerium S. de R.L. de C.V., Monterrey
  - Hospital Universitario Dr Jose Eleuterio Gonzalez; Universidad Autónoma de Nuevo León, Monterrey
- Poland (15):
  - Centrum Medyczne Sw. Lukasza, Częstochowa
  - 7 Szpital Marynarki Wojennej z Przychodnia SPZOZ im. W. Lasinskiego, Gdansk
  - NZOZ Centrum Medyczne ProMiMed, Krakow
  - AppleTreeClinics Sp. z o.o., Lodz
  - Med-Gastr Przychodnia Specjalistyczna, Lodz
  - Indywidualna Specjalistyczna Praktyka Lekarska, Lublin
  - GASTROMED Sp. z o.o., Lublin
  - Wojewodzki Specjalistyczny Szpital w Olsztynie, Olsztyn
  - SOLUMED Centrum Medyczne, Poznan
  - Specjalistyczna Praktyka Lekarska Dr med. Marek Horynski; endoskopia, Sopot
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
  - EMC Instytut Medyczny S.A., Wroclaw
  - PlanetMed, Wroclaw
- Russia (14):
  - Yusupov Hospital, Moskva, Adygeya Republic
  - SPb SBIH "City Multy-field Hospital # 2"; Intensive Pulmonology and Thoracal Surgery, Saint Petersburg, Sankt-Peterburg
  - Baltic Medicine, Saint Petersburg, Sankt-Peterburg
  - Medical and Sanitary Division of Severstal, Cherepovets, Vologda Oblast
  - SBEI HPE Altai State Medical University of MoH and SD; Out-patient Department, Barnaul
  - FSBIH Central Clinical Hospital of RAS, Moscow
  - FSBI "State Scientific Centre of Coloproctology" of the MoH of RF; Gastroenterology, Moscow
  - SBHI of NN region "RCH of NN n.a. N.A.Semashko", Nizhny Novgorod
  - SBEI of HPE "Omsk SMA" Ministry of healthcare of RF", Omsk
  - SEIHPE "Rostov SMU of MoH of RF", Rostov-on-Don
  - FSMEI HPE "Military Medical Academy n.a. S.M.Kirov"of Minist, Saint Petersburg
  - City Hospital #26, Saint Petersburg
  - LLC International Medical Centre "SOGAZ", Saint Petersburg
  - Stavropol Regional Clinical Diagnostic Consultative Center, Stavropol
- Serbia (6):
  - Clinical Center Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
  - Clinical Center Zemun, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - General Hospital "Djordje Joanovic"; Gastroenterology, Zrenjanin
- Slovakia (6):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Nemocnica A.Lena Humenne, n.o., Humenné
  - KM Management spol. s r.o., Nitra
  - Gastro I, s.r.o., Prešov
  - Svet zdravia a.s., Rimavská Sobota
  - Accout Center s.r.o., Šahy
- Ukraine (11):
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2 of KCC, Kharkiv, Kharkiv Governorate
  - Communal Non-commercial Enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv, Kharkiv Governorate
  - Communal Institution of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv, Kharkiv Governorate
  - Medical Center of Limited Liability Company Medical Clinic Blagomed, Kyiv, KIEV Governorate
  - CI of Kyiv RC Regional Clinical Hospital #2, Kyiv, KIEV Governorate
  - CI City Hospital #1, Zaporizhzhia, Tavria Okruha
  - RCI Chernivtsi RCH Gastroenterology Bukovinsky SMU, Chernivtsi
  - CHI Kharkiv City Clinical Hospital #13, Kharkiv
  - CNI Consultative and Diagnostic Center of Desnianskyi District of Kyiv, Kyiv
  - M.V. Sklifosovskyi Poltava RCH Outpatient UMSA HSEIU Ukrainian Medical Stomatological Academy, Poltava
  - CI City Hospital #7, Zaporizhzhia

REFERENCES:
- [Derived] Rubin DT, Dotan I, DuVall A, Bouhnik Y, Radford-Smith G, Higgins PDR, Mishkin DS, Arrisi P, Scalori A, Oh YS, Tole S, Chai A, Chamberlain-James K, Lacey S, McBride J, Panes J; HIBISCUS Study Group. Etrolizumab versus adalimumab or placebo as induction therapy for moderately to severely active ulcerative colitis (HIBISCUS): two phase 3 randomised, controlled trials. Lancet Gastroenterol Hepatol. 2022 Jan;7(1):17-27. doi: 10.1016/S2468-1253(21)00338-1. Epub 2021 Nov 17. PMID 34798036
- [Derived] Sandborn WJ, Vermeire S, Tyrrell H, Hassanali A, Lacey S, Tole S, Tatro AR; Etrolizumab Global Steering Committee. Etrolizumab for the Treatment of Ulcerative Colitis and Crohn's Disease: An Overview of the Phase 3 Clinical Program. Adv Ther. 2020 Jul;37(7):3417-3431. doi: 10.1007/s12325-020-01366-2. Epub 2020 May 22. PMID 32445184

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were on concomitant background therapy were allowed to continue receiving stable baseline doses of the following non-investigational medicinal products during the study: oral 5-aminosalicylic acid; azathioprine; 6-mercaptopurine; methotrexate; corticosteroids up to 30 mg/day of prednisone (or equivalent); and/or budesonide up to 9 mg/day.
Groups:
- Placebo: The double-blinded treatment period consisted of a 10-week induction period and an additional 4-week treatment period for participants who met the definition of clinical remission at Week 10. Participants with moderate-to-severe ulcerative colitis who were naive to TNF inhibitors were randomized to this arm to receive placebo matching to etrolizumab subcutaneously (SC) once every 4 weeks (Q4W) up to Week 12 (at Weeks 0 [Day 1], 4, 8, and 12 [clinical remitters only]) and placebo matching to adalimumab SC once every 2 weeks (Q2W) up to Week 8 (at Weeks 0 [Day 1], 2, 4, 6, and 8).
- Adalimumab: The double-blinded treatment period consisted of a 10-week induction period and an additional 4-week treatment period for participants who met the definition of clinical remission at Week 10. Participants with moderate-to-severe ulcerative colitis who were naive to TNF inhibitors were randomized to this arm to receive adalimumab subcutaneously (SC) Q2W up to Week 8 (160 mg at Week 0 [Day 1], 80 mg at Week 2, 40 mg at Weeks 4, 6, and 8) and placebo matching to etrolizumab SC Q4W up to Week 12 (at Weeks 0 [Day 1], 4, 8, and 12 [clinical remitters only]).
- Etrolizumab: The double-blinded treatment period consisted of a 10-week induction period and an additional 4-week treatment period for participants who met the definition of clinical remission at Week 10. Participants with moderate-to-severe ulcerative colitis who were naive to TNF inhibitors were randomized to this arm to receive etrolizumab 105 mg subcutaneously (SC) Q4W up to Week 12 (at Weeks 0 [Day 1], 4, 8, and 12 [clinical remitters only]) and placebo matching to adalimumab SC Q2W up to Week 8 (at Weeks 0 [Day 1], 2, 4, 6, and 8).
Period: Overall Study
Arm/Group | Placebo | Adalimumab | Etrolizumab
Started | 72 | 142 | 144
Completed Week 10 | 71 | 141 | 143
Completed (Participants who rolled into open-label extension study or completed 12 weeks safety follow-up following treatment completion or discontinuation.) | 71 | 137 | 141
Not Completed | 1 | 5 | 3
Not completed — Withdrawal by Subject | 1 | 5 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants (716) represents the total number enrolled (358) in this study, GA28948 (NCT02163759), plus the total number enrolled (358) in a second study of identical design, GA28949 (NCT02171429). Some of the pre-specified secondary outcome measure comparisons were planned to be evaluated by pooling data from both studies; all etrolizumab versus adalimumab comparisons and one family of etrolizumab versus placebo comparisons were evaluated on pooled data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab | Etrolizumab | Total
Number analyzed (Participants) | 144 | 285 | 287 | 716
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Baseline characteristics are presented for two populations: all 358 participants enrolled in this study, GA28948 (NCT02163759); and a total pooled population of 716 participants, which consists of all 358 participants from this study (GA28948) plus all 358 participants enrolled in a second study of identical design, GA28949 (NCT02171429).
  Years
    GA28948 Population: number analyzed (Participants) | 72 | 142 | 144 | 358
    GA28948 Population | 38.4 (13.3) | 42.0 (13.8) | 40.1 (13.4) | 40.5 (13.5)
    GA28948 & GA28949 Pooled Population | 39.4 (12.9) | 40.8 (13.2) | 40.6 (13.9) | 40.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics are presented for two populations: all 358 participants enrolled in this study, GA28948 (NCT02163759); and a total pooled population of 716 participants, which consists of all 358 participants from this study (GA28948) plus all 358 participants enrolled in a second study of identical design, GA28949 (NCT02171429).
  Participants
    GA28948 Population: number analyzed (Participants) | 72 | 142 | 144 | 358
    GA28948 Population: Female | 33 | 60 | 70 | 163
    GA28948 Population: Male | 39 | 82 | 74 | 195
    GA28948 & GA28949 Pooled Population: Female | 67 | 122 | 129 | 318
    GA28948 & GA28949 Pooled Population: Male | 77 | 163 | 158 | 398
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics are presented for two populations: all 358 participants enrolled in this study, GA28948 (NCT02163759); and a total pooled population of 716 participants, which consists of all 358 participants from this study (GA28948) plus all 358 participants enrolled in a second study of identical design, GA28949 (NCT02171429).
  Participants
    GA28948 Population: number analyzed (Participants) | 72 | 142 | 144 | 358
    GA28948 Population: Hispanic or Latino | 8 | 16 | 14 | 38
    GA28948 Population: Not Hispanic or Latino | 63 | 123 | 128 | 314
    GA28948 Population: Unknown or Not Reported | 1 | 3 | 2 | 6
    GA28948 & GA28949 Pooled Population: Hispanic or Latino | 13 | 27 | 26 | 66
    GA28948 & GA28949 Pooled Population: Not Hispanic or Latino | 130 | 253 | 256 | 639
    GA28948 & GA28949 Pooled Population: Unknown or Not Reported | 1 | 5 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics are presented for two populations: all 358 participants enrolled in this study, GA28948 (NCT02163759); and a total pooled population of 716 participants, which consists of all 358 participants from this study (GA28948) plus all 358 participants enrolled in a second study of identical design, GA28949 (NCT02171429).
  Participants
    GA28948 Population: number analyzed (Participants) | 72 | 142 | 144 | 358
    GA28948 Population: Asian | 0 | 2 | 0 | 2
    GA28948 Population: Black or African American | 2 | 0 | 1 | 3
    GA28948 Population: White | 68 | 130 | 138 | 336
    GA28948 Population: Other | 2 | 10 | 5 | 17
    GA28948 & GA28949 Pooled Population: Asian | 4 | 6 | 4 | 14
    GA28948 & GA28949 Pooled Population: Black or African American | 3 | 4 | 2 | 9
    GA28948 & GA28949 Pooled Population: White | 133 | 261 | 271 | 665
    GA28948 & GA28949 Pooled Population: Other | 4 | 14 | 10 | 28
Disease Location [Count of Participants; unit: Participants] — Population: Baseline characteristics are presented for two populations: all 358 participants enrolled in this study, GA28948 (NCT02163759); and a total pooled population of 716 participants, which consists of all 358 participants from this study (GA28948) plus all 358 participants enrolled in a second study of identical design, GA28949 (NCT02171429).
  Participants
    GA28948 Population: number analyzed (Participants) | 72 | 142 | 144 | 358
    GA28948 Population: Left-Sided Colitis | 44 | 84 | 89 | 217
    GA28948 Population: Extensive Colitis | 10 | 23 | 22 | 55
    GA28948 Population: Pancolitis | 18 | 35 | 33 | 86
    GA28948 & GA28949 Pooled Population: Left-Sided Colitis | 92 | 170 | 175 | 437
    GA28948 & GA28949 Pooled Population: Extensive Colitis | 17 | 36 | 33 | 86
    GA28948 & GA28949 Pooled Population: Pancolitis | 35 | 79 | 79 | 193
Mayo Clinic Score (MCS) ≤9 or ≥10 at Baseline [Count of Participants; unit: Participants] — Participants were stratified by concomitant treatment with corticosteroids (yes/no) at randomization, concomitant treatment with immunosuppressants (yes/no) at randomization, and disease activity measured during screening (MCS ≤9/MCS ≥10). The MCS ranges from 0 to 12 and is a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and physician's global assessment (PGA) subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease. Population: Baseline characteristics are presented for two populations: all 358 participants enrolled in this study, GA28948 (NCT02163759); and a total pooled population of 716 participants, which consists of all 358 participants from this study (GA28948) plus all 358 participants enrolled in a second study of identical design, GA28949 (NCT02171429).
  Participants
    GA28948 Population: number analyzed (Participants) | 72 | 142 | 144 | 358
    GA28948 Population: MCS ≤9 | 47 | 96 | 100 | 243
    GA28948 Population: MCS ≥10 | 25 | 46 | 44 | 115
    GA28948 & GA28949 Pooled Population: MCS ≤9 | 93 | 192 | 196 | 481
    GA28948 & GA28949 Pooled Population: MCS ≥10 | 51 | 93 | 91 | 235
Baseline Treatment: None, Corticosteroids (CS) or Immunosuppressants (IS) Alone, or Both CS and IS [Count of Participants; unit: Participants] — Participants were stratified by concomitant treatment with corticosteroids (yes/no) at randomization, concomitant treatment with immunosuppressants (yes/no) at randomization, and disease activity measured during screening (MCS ≤9/MCS ≥10). Population: Baseline characteristics are presented for two populations: all 358 participants enrolled in this study, GA28948 (NCT02163759); and a total pooled population of 716 participants, which consists of all 358 participants from this study (GA28948) plus all 358 participants enrolled in a second study of identical design, GA28949 (NCT02171429).
  Participants
    GA28948 Population: number analyzed (Participants) | 72 | 142 | 144 | 358
    GA28948 Population: None | 24 | 51 | 45 | 120
    GA28948 Population: Corticosteroids (CS) Alone | 25 | 46 | 50 | 121
    GA28948 Population: Immunosuppressants (IS) Alone | 15 | 30 | 32 | 77
    GA28948 Population: Both CS and IS | 8 | 15 | 17 | 40
    GA28948 & GA28949 Pooled Population: None | 51 | 104 | 100 | 255
    GA28948 & GA28949 Pooled Population: Corticosteroids (CS) Alone | 48 | 88 | 90 | 226
    GA28948 & GA28949 Pooled Population: Immunosuppressants (IS) Alone | 29 | 58 | 60 | 147
    GA28948 & GA28949 Pooled Population: Both CS and IS | 16 | 35 | 37 | 88
Nancy Histological Index (NHI) Score of ≤1 or >1, or Missing, at Baseline [Count of Participants; unit: Participants] — Histologic disease activity was measured using the Nancy Histological Index (NHI) score, ranging from 0 to 4, with the following definitions for each grade: 0 is no histologically significant disease; 1 is chronic inflammatory infiltrate with no acute inflammatory infiltrate; and 2, 3, and 4 are mildly, moderately, and severely active disease, respectively. Population: Baseline characteristics are presented for two populations: all 358 participants enrolled in this study, GA28948 (NCT02163759); and a total pooled population of 716 participants, which consists of all 358 participants from this study (GA28948) plus all 358 participants enrolled in a second study of identical design, GA28949 (NCT02171429).
  Participants
    GA28948 Population: number analyzed (Participants) | 72 | 142 | 144 | 358
    GA28948 Population: NHI Score ≤1 | 8 | 15 | 15 | 38
    GA28948 Population: NHI Score >1 | 62 | 116 | 120 | 298
    GA28948 Population: Missing | 2 | 11 | 9 | 22
    GA28948 & GA28949 Pooled Population: NHI Score ≤1 | 17 | 38 | 36 | 91
    GA28948 & GA28949 Pooled Population: NHI Score >1 | 124 | 230 | 228 | 582
    GA28948 & GA28949 Pooled Population: Missing | 3 | 17 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Remission at Week 10 With Etrolizumab as Compared With Placebo, as Determined by the Mayo Clinic Score (MCS), GA28948 Population
Description: The Mayo Clinic Score (MCS) ranges from 0 to 12 and is a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and physician's global assessment (PGA) subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease. Remission was defined as MCS less than or equal to (≤)2 with individual subscores ≤1 and a rectal bleeding subscore of 0. Participants were also classified as non-remitters if Week 10 assessments were missing or if they had received permitted/prohibited rescue therapy prior to assessment. Participants were stratified by concomitant treatment with corticosteroids or immunosuppressants at randomization and disease activity measured during screening (MCS ≤9/MCS ≥10); the Cochran-Mantel-Haenszel test adjusted the difference in remission rates and associated 95% confidence interval for the stratification factors.
Time Frame: Week 10
Population: GA28948 Population, Modified Intent-to-Treat: including all randomized participants in study GA28948 who received at least one dose of study drug, with participants grouped according to the treatment assigned at randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Etrolizumab
Number analyzed (Participants) | 72 | 144
Percentage of participants | 6.9 [3.00 to 15.25] | 19.4 [13.81 to 26.67]
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; The null hypothesis (H0): the percentage of participants achieving remission at Week 10 was the same in both the placebo and etrolizumab arms. The alternative hypothesis (H1): the percentage of participants achieving remission at Week 10 was not the same in the placebo and etrolizumab arms; Test type: Superiority; p = 0.0173, Cochran-Mantel-Haenszel — The threshold for statistical significance was a p-value <0.05; Difference and 95% CI adjusted for concomitant treatment with corticosteroids or immunosuppressants at baseline (BL) and MCS (≤9 or ≥10) at BL; Difference in Remission Rates = 12.3, 95% CI 2-sided [1.59 to 20.60] — Difference in remission rates was calculated as the etrolizumab arm minus the placebo arm

2. Secondary Outcome: Percentage of Participants in Remission at Week 10 With Etrolizumab as Compared With Adalimumab, as Determined by the MCS, GA28948 Population
Description: The Mayo Clinic Score (MCS) ranges from 0 to 12 and is a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and physician's global assessment (PGA) subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease. Remission was defined as MCS less than or equal to (≤)2 with individual subscores ≤1 and a rectal bleeding subscore of 0. Participants were also classified as non-remitters if Week 10 assessments were missing or if they had received permitted/prohibited rescue therapy prior to assessment. Participants were stratified by concomitant treatment with corticosteroids or immunosuppressants at randomization and disease activity measured during screening (MCS ≤9/MCS ≥10). The Cochran-Mantel-Haenszel test adjusted the difference in remission rates and associated 95% confidence interval for the stratification factors.
Time Frame: Week 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adalimumab | Etrolizumab
Number analyzed (Participants) | 142 | 144
Percentage of participants | 22.5 [16.44 to 30.08] | 19.4 [13.81 to 26.67]
Statistical Analysis 1: Comparison: Adalimumab vs Etrolizumab; Primary and secondary outcome measures were evaluated for statistical significance in a hierarchical manner with a component-wise multistage gatekeeping procedure. Please refer to the statistical analysis plan for details. This comparison was not considered a key secondary outcome measure and was not part of the multiple testing procedure for statistical significance; Test type: Superiority; p = 0.5055, Cochran-Mantel-Haenszel — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = -3.1, 95% CI 2-sided [-12.61 to 6.37] — Difference in remission rates was calculated as the etrolizumab arm minus the adalimumab arm

3. Secondary Outcome: Percentage of Participants in Remission at Week 10 With Etrolizumab as Compared With Adalimumab, as Determined by the MCS, GA28948 & GA28949 Pooled Population
Description: as for outcome 2
Time Frame: Week 10
Population: GA28948 & GA28949 Pooled Population, Modified Intent-to-Treat: including all randomized participants in studies GA28948 & GA28949 who received at least one dose of study drug, with participants grouped according to the treatment assigned at randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adalimumab | Etrolizumab
Number analyzed (Participants) | 285 | 287
Percentage of participants | 23.5 [18.96 to 28.76] | 18.8 [14.72 to 23.74]
Statistical Analysis 1: Comparison: Adalimumab vs Etrolizumab; Primary and secondary outcome measures were evaluated for statistical significance in a hierarchical manner with a component-wise multistage gatekeeping procedure. This comparison was part of Family 3 of the testing procedure; please refer to the statistical analysis plan for details; Test type: Superiority; p = 1, Cochran-Mantel-Haenszel — p-value has been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = -5.0, 95% CI 2-sided [-11.66 to 1.75] — Difference in remission rates was calculated as the etrolizumab arm minus the adalimumab arm

4. Secondary Outcome: Percentage of Participants With Clinical Response at Week 10, as Determined by the MCS, GA28948 Population
Description: The Mayo Clinic Score (MCS) ranges from 0 to 12 and is a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and physician's global assessment subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease. Clinical Response was defined as: MCS ≥3-point decrease and 30% reduction from baseline as well as ≥1-point decrease in rectal bleeding subscore or an absolute rectal bleeding score of 0 or 1. Non-responders also included participants with missing Week 10 assessments or those who had received permitted/prohibited rescue therapy prior to assessment. Participants were stratified by concomitant treatment with corticosteroids or immunosuppressants at randomization and disease activity measured during screening (MCS ≤9 or ≥10); the CMH test adjusted the differences in response rates and associated 95% CIs for the stratification factors.
Time Frame: Week 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 72 | 142 | 144
Percentage of participants | 50.0 [38.75 to 61.25] | 52.1 [43.95 to 60.16] | 56.9 [48.78 to 64.75]
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; Primary and secondary outcome measures were evaluated for statistical significance in a hierarchical manner with a component-wise multistage gatekeeping procedure. This comparison was part of Family 1 of the testing procedure; please refer to the statistical analysis plan for details; Test type: Superiority; p = 0.4434, Cochran-Mantel-Haenszel — p-value has been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Response Rates = 6.9, 95% CI 2-sided [-7.03 to 20.62] — Difference in response rates was calculated as the etrolizumab arm minus the placebo arm
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4122, Cochran-Mantel-Haenszel — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Response Rates = 4.8, 95% CI 2-sided [-6.72 to 16.07] — Difference in response rates was calculated as the etrolizumab arm minus the adalimumab arm

5. Secondary Outcome: Percentage of Participants With Clinical Response at Week 10 With Etrolizumab as Compared With Adalimumab, as Determined by the MCS, GA28948 & GA28949 Pooled Population
Description: as for outcome 4
Time Frame: Week 10
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adalimumab | Etrolizumab
Number analyzed (Participants) | 285 | 287
Percentage of participants | 53.3 [47.54 to 59.04] | 54.7 [48.92 to 60.36]
Statistical Analysis 1: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 1, Cochran-Mantel-Haenszel — p-value has been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Response Rates = 1.2, 95% CI 2-sided [-6.98 to 9.26] — Difference in response rates was calculated as the etrolizumab arm minus the adalimumab arm

6. Secondary Outcome: Percentage of Participants With Improvement in Endoscopic Appearance of the Mucosa at Week 10, as Determined by the MCS Endoscopy Subscore, GA28948 Population
Description: Improvement in endoscopic appearance of the mucosa was defined as a Mayo Clinic Score (MCS) endoscopy subscore ≤1. Blinded gastroenterologists experienced in inflammatory bowel disease performed central reading of endoscopies at an independent review facility. The rectum, sigmoid, and descending colon segments were assessed and each segment was assigned a score of 0 to 3, with higher scores indicating more severe disease. At baseline all segments were reviewed and the worst score from the three segments was recorded as the endoscopy subscore. Post-baseline the endoscopy score was the worst score of all segments that had been assessed at baseline, if the baseline endoscopy score had a sigmoid colon score ≤1. If at baseline the sigmoid colon score was ≥2, the post-baseline endoscopy score was the sigmoid colon score value. Non-responders also included participants with missing Week 10 assessments or those who had received permitted/prohibited rescue therapy prior to assessment.
Time Frame: Week 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 72 | 142 | 144
Percentage of participants | 22.2 [14.17 to 33.09] | 33.1 [25.89 to 41.19] | 40.3 [32.62 to 48.44]
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0173, Cochran-Mantel-Haenszel — p-value has been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Response Rates = 17.9, 95% CI 2-sided [4.49 to 29.50] — Difference in response rates was calculated as the etrolizumab arm minus the placebo arm
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1886, Cochran-Mantel-Haenszel — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Response Rates = 7.4, 95% CI 2-sided [-3.77 to 18.32] — Difference in response rates was calculated as the etrolizumab arm minus the adalimumab arm

7. Secondary Outcome: Percentage of Participants With Improvement in Endoscopic Appearance of the Mucosa at Week 10 With Etrolizumab as Compared With Adalimumab, as Determined by the MCS Endoscopy Subscore, GA28948 & GA28949 Pooled Population
Description: as for outcome 6
Time Frame: Week 10
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adalimumab | Etrolizumab
Number analyzed (Participants) | 285 | 287
Percentage of participants | 37.9 [32.46 to 43.65] | 40.1 [34.57 to 45.83]
Statistical Analysis 1: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 1, Cochran-Mantel-Haenszel — p-value has been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Response Rates = 1.9, 95% CI 2-sided [-6.04 to 9.88] — Difference in response rates was calculated as the etrolizumab arm minus the adalimumab arm

8. Secondary Outcome: Percentage of Participants in Endoscopic Remission at Week 10, as Determined by the MCS Endoscopy Subscore, GA28948 Population
Description: Endoscopic remission was defined as a Mayo Clinic Score (MCS) endoscopy subscore of 0. Blinded gastroenterologists experienced in inflammatory bowel disease performed central reading of endoscopies at an independent review facility. The rectum, sigmoid, and descending colon segments were assessed and each segment was assigned a score of 0 to 3, with higher scores indicating more severe disease. At baseline all segments were reviewed and the worst score from the three segments was recorded as the endoscopy subscore. Post-baseline the endoscopy score was the worst score of all segments that had been assessed at baseline, if the baseline endoscopy score had a sigmoid colon score ≤1. If at baseline the sigmoid colon score was ≥2, the post-baseline endoscopy score was the sigmoid colon score value. Non-responders also included participants with missing Week 10 assessments or those who had received permitted/prohibited rescue therapy prior to assessment.
Time Frame: Week 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 72 | 142 | 144
Percentage of participants | 6.9 [3.00 to 15.25] | 20.4 [14.61 to 27.79] | 20.8 [15.00 to 28.18]
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; Primary and secondary outcome measures were evaluated for statistical significance in a hierarchical manner with a component-wise multistage gatekeeping procedure. This comparison was part of Family 2 of the testing procedure; please refer to the statistical analysis plan for details; Test type: Superiority; p = 0.1347, Cochran-Mantel-Haenszel — p-value has been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = 13.8, 95% CI 2-sided [2.97 to 22.15] — Difference in remission rates was calculated as the etrolizumab arm minus the placebo arm
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9138, Cochran-Mantel-Haenszel — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = 0.5, 95% CI 2-sided [-8.95 to 9.92] — Difference in remission rates was calculated as the etrolizumab arm minus the adalimumab arm

9. Secondary Outcome: Percentage of Participants in Endoscopic Remission at Week 10 With Etrolizumab as Compared With Adalimumab, as Determined by the MCS Endoscopy Subscore, GA28948 & GA28949 Pooled Population
Description: as for outcome 8
Time Frame: Week 10
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adalimumab | Etrolizumab
Number analyzed (Participants) | 285 | 287
Percentage of participants | 23.5 [18.96 to 28.76] | 20.2 [15.97 to 25.23]
Statistical Analysis 1: Comparison: Adalimumab vs Etrolizumab; Primary and secondary outcome measures were evaluated for statistical significance in a hierarchical manner with a component-wise multistage gatekeeping procedure. This comparison was part of Family 5 of the testing procedure; please refer to the statistical analysis plan for details; Test type: Superiority; p = 1, Cochran-Mantel-Haenszel — p-value has been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = -3.5, 95% CI 2-sided [-10.27 to 3.30] — Difference in remission rates was calculated as the etrolizumab arm minus the adalimumab arm

10. Secondary Outcome: Percentage of Participants With Histologic Remission at Week 10, as Determined by the Nancy Histological Index, GA28948 Population
Description: Histologic remission is defined by the resolution of neutrophilic inflammation (e.g., absence of neutrophils in the crypts and lamina propria), defined by a Nancy Histological Index (NHI) score of ≤1. The NHI score ranges from 0 to 4, with the following definitions for each grade: 0 is no histologically significant disease; 1 is chronic inflammatory infiltrate with no acute inflammatory infiltrate; and 2, 3, and 4 are mildly, moderately, and severely active disease, respectively. A small pool of central readers who were blinded to both treatment arm and timepoint performed the histologic scoring. The same reader scored all slides for a given participant based on biopsies from the most inflamed region of the sigmoid colon. Participants were also classified as non-remitters if Week 10 assessments were missing or if they had received rescue therapy prior to assessment. The Cochran-Mantel-Haenszel test adjusted the difference in remission rates and 95% CI for the stratification factors.
Time Frame: Week 10
Population: GA28948 Histology-Evaluable Population: included all randomized participants in study GA28948 who received at least one dose of study drug and had documented neutrophilic inflammation (i.e., NHI >1) at baseline. This excludes participants who had no baseline histology assessment or had no indication of neutrophilic inflammation at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 62 | 116 | 120
Percentage of participants | 16.1 [9.00 to 27.21] | 29.3 [21.80 to 38.15] | 42.5 [34.02 to 51.44]
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0173, Cochran-Mantel-Haenszel — p-value has been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = 26.3, 95% CI 2-sided [12.10 to 37.86] — Difference in remission rates was calculated as the etrolizumab arm minus the placebo arm
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0313, Cochran-Mantel-Haenszel — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = 13.2, 95% CI 2-sided [0.93 to 24.94] — Difference in remission rates was calculated as the etrolizumab arm minus the adalimumab arm

11. Secondary Outcome: Percentage of Participants With Histologic Remission at Week 10 With Etrolizumab as Compared With Adalimumab, as Determined by the Nancy Histological Index, GA28948 & GA28949 Pooled Population
Description: as for outcome 10
Time Frame: Week 10
Population: GA28948 & GA28949 Pooled, Histology-Evaluable Population: included all randomized participants in studies GA28948 & GA28949 who received at least one dose of study drug and had documented neutrophilic inflammation (i.e., NHI >1) at baseline. This excludes participants who had no baseline histology assessment or had no indication of neutrophilic inflammation at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Adalimumab | Etrolizumab
Number analyzed (Participants) | 230 | 228
Percentage of participants | 36.5 [30.57 to 42.92] | 36.8 [30.85 to 43.27]
Statistical Analysis 1: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 1, Cochran-Mantel-Haenszel — p-value has been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = -0.3, 95% CI 2-sided [-9.13 to 8.45] — Difference in remission rates was calculated as the etrolizumab arm minus the adalimumab arm

12. Secondary Outcome: Change From Baseline in the MCS Rectal Bleeding Subscore at Week 6, GA28948 Population
Description: Rectal bleeding data were collected via the participant's diaries and each day a participant provided a score from 0 to 3 according to the following definitions: 0 = no blood in the stool; 1 = streaks of blood with stool less than half the time; 2 = obvious blood with stool most of the time; 3 = blood alone passed. The Mayo Clinic Score (MCS) rectal bleeding subscore was calculated as the worst value of three days of daily diary scores closest to anchor dates at baseline and post-baseline. The data was considered non-parametric and was reported using RANK analysis of covariance (ANCOVA). Participants were stratified by concomitant treatment with corticosteroids or immunosuppressants at randomization and disease activity measured during screening (MCS ≤9/MCS ≥10); the model adjusted for these stratification factors along with the baseline rectal bleeding (RB) subscore.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 72 | 142 | 144
Score on a scale | -1.0 [-1.0 to 0.0] | -1.0 [-2.0 to 0.0] | -1.0 [-2.0 to 0.0]
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.4434, Rank ANCOVA — p-value has been adjusted for multiplicity; Model adjusted for concomitant treatment with corticosteroids or immunosuppressants at baseline (BL), MCS (≤9 or ≥10) at BL, and RB score at BL
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3374, Rank ANCOVA — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 12, analysis 1]

13. Secondary Outcome: Change From Baseline in the MCS Rectal Bleeding Subscore at Week 6 With Etrolizumab as Compared With Adalimumab, GA28948 & GA28949 Pooled Population
Description: as for outcome 12
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Adalimumab | Etrolizumab
Number analyzed (Participants) | 285 | 287
Score on a scale | -1.0 [-2.0 to 0.0] | -1.0 [-2.0 to 0.0]
Statistical Analysis 1: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 1, Rank ANCOVA — p-value has been adjusted for multiplicity; [statistical method as in outcome 12, analysis 1]

14. Secondary Outcome: Change From Baseline in the MCS Stool Frequency Subscore at Week 6, GA28948 Population
Description: Stool frequency data were collected via the participant's diaries and each day a participant provided a score from 0 to 3 according to the following definitions: 0 = normal number of stools; 1 = 1 to 2 more stools than normal; 2 = 3 to 4 more stools than normal; 3 = 5 or more stools than normal. The Mayo Clinic Score (MCS) stool frequency subscore was calculated as the average of three days daily diary scores closest to anchor dates at baseline and post-baseline. The data was considered non-parametric and was reported using RANK analysis of covariance (ANCOVA). Participants were stratified by concomitant treatment with corticosteroids or immunosuppressants at randomization and disease activity measured during screening (MCS ≤9/MCS ≥10); the model adjusted for these stratification factors along with the baseline stool frequency (SF) subscore.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 72 | 142 | 144
Score on a scale | 0.0 [-1.0 to 0.0] | -1.0 [-2.0 to 0.0] | -1.0 [-2.0 to 0.0]
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.4434, Rank ANCOVA — p-value has been adjusted for multiplicity; Model adjusted for concomitant treatment with corticosteroids or immunosuppressants at baseline (BL), MCS (≤9 or ≥10) at BL, and SF score at BL
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6367, Rank ANCOVA — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 14, analysis 1]

15. Secondary Outcome: Change From Baseline in the MCS Stool Frequency Subscore at Week 6 With Etrolizumab as Compared With Adalimumab, GA28948 & GA28949 Pooled Population
Description: as for outcome 14
Time Frame: Baseline, Week 6
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Adalimumab | Etrolizumab
Number analyzed (Participants) | 285 | 287
Score on a scale | -1.0 [-1.0 to 0.0] | -1.0 [-1.0 to 0.0]
Statistical Analysis 1: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 1, Rank ANCOVA — p-value has been adjusted for multiplicity; [statistical method as in outcome 14, analysis 1]

16. Secondary Outcome: Change From Baseline in Ulcerative Colitis (UC) Bowel Movement Signs and Symptoms at Week 10, as Assessed by the UC Patient-Reported Outcome Signs and Symptoms (UC-PRO/SS), GA28948 Population
Description: The UC-PRO/SS questionnaire was collected in the e-diary and completed by participants for at least 9 to 12 consecutive days prior to a study visit. The bowel movement domain score ranges from 0 to 27, with a higher score indicating a worse disease state. The most recent 7 daily scores available (not including the visit) were selected for the calculation of the visit score. For each item in the questionnaire, a score was calculated for a visit by taking the average of the selected daily scores. The domain score for a visit was calculated as the sum of the averaged items for each question. A Mixed Model for Repeated Measures (MMRM) analysis of the data included the fixed categorical effects of treatment, visit, study stratification factors, and treatment-by-visit interaction, and the continuous covariates of the baseline UC-PRO/SS domain and baseline UC-PRO/SS domain-by-visit interaction. An unstructured covariance matrix was used to model the within-patient errors within the MMRM.
Time Frame: Baseline, Week 10
Population: GA28948 Population, Modified Intent-to-Treat: including all randomized participants in study GA28948 who received at least one dose of study drug, with participants grouped according to the treatment assigned at randomization. The analysis only included participants with non-missing results at baseline and at least one post-baseline timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 50 | 106 | 117
Score on a scale | -5.5 (0.7) | -5.7 (0.5) | -6.2 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3708, Mixed Model for Repeated Measures — Nominal p-value; it has not been adjusted for multiplicity; Model adjusted for treatment, visit, stratification factors, treatment-by-visit, baseline UC-PRO/SS domain, and baseline UC-PRO/SS domain-by-visit; Mean Difference (Net) = -0.7, 95% CI 2-sided [-2.4 to 0.9] — Mean difference was calculated as etrolizumab arm minus placebo arm
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4477, Mixed Model for Repeated Measures — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 16, analysis 1]; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.8 to 0.8] — Mean difference was calculated as etrolizumab arm minus adalimumab arm

17. Secondary Outcome: Change From Baseline in Ulcerative Colitis Bowel Movement Signs and Symptoms at Week 10, as Assessed by the UC-PRO/SS, GA28948 & GA28949 Pooled Population
Description: as for outcome 16
Time Frame: Baseline, Week 10
Population: GA28948 & GA28949 Pooled Population, Modified Intent-to-Treat: including all randomized participants in studies GA28948 & GA28949 who received at least one dose of study drug, with participants grouped according to the treatment assigned at randomization. The analysis only included participants with non-missing results at baseline and at least one post-baseline timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 109 | 217 | 225
Score on a scale | -5.0 (0.5) | -5.8 (0.4) | -6.0 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; Primary and secondary outcome measures were evaluated for statistical significance in a hierarchical manner with a component-wise multistage gatekeeping procedure. This comparison was part of Family 4 of the testing procedure; please refer to the statistical analysis plan for details; Test type: Superiority; p = 1, Mixed Model for Repeated Measures — p-value has been adjusted for multiplicity; [statistical method as in outcome 16, analysis 1]; Mean Difference (Net) = -1.0, 95% CI 2-sided [-2.1 to 0.2] — Mean difference was calculated as etrolizumab arm minus placebo arm
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; Primary and secondary outcome measures were evaluated for statistical significance in a hierarchical manner with a component-wise multistage gatekeeping procedure. This comparison was part of Family 6 of the testing procedure; please refer to the statistical analysis plan for details; Test type: Superiority; p = 1, Mixed Model for Repeated Measures — p-value has been adjusted for multiplicity; [statistical method as in outcome 16, analysis 1]; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.2 to 0.7] — Mean difference was calculated as etrolizumab arm minus adalimumab arm

18. Secondary Outcome: Change From Baseline in Ulcerative Colitis Functional Symptoms at Week 10, as Assessed by the UC-PRO/SS, GA28948 Population
Description: The UC-PRO/SS questionnaire was collected in the e-diary and completed by participants for at least 9 to 12 consecutive days prior to a study visit. The functional symptoms domain score ranges from 0 to 12, with a higher score indicating a worse disease state. The most recent 7 daily scores available (not including the visit) were selected for the calculation of the visit score. For each item in the questionnaire, a score was calculated for a visit by taking the average of the selected daily scores. The domain score for a visit was calculated as the sum of the averaged items for each question. A Mixed Model for Repeated Measures (MMRM) analysis of the data included the fixed categorical effects of treatment, visit, study stratification factors, and treatment-by-visit interaction, and the continuous covariates of the baseline UC-PRO/SS domain and baseline UC-PRO/SS domain-by-visit interaction. An unstructured covariance matrix was used to model the within-patient errors in the MMRM.
Time Frame: Baseline, Week 10
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 50 | 106 | 117
Score on a scale | -1.7 (0.3) | -1.5 (0.2) | -1.9 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6356, Mixed Model for Repeated Measures — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 16, analysis 1]; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.9 to 0.5] — Mean difference was calculated as etrolizumab arm minus placebo arm
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1253, Mixed Model for Repeated Measures — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 16, analysis 1]; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.0 to 0.1] — Mean difference was calculated as etrolizumab arm minus adalimumab arm

19. Secondary Outcome: Change From Baseline in Ulcerative Colitis Functional Symptoms at Week 10, as Assessed by the UC-PRO/SS, GA28948 & GA28949 Pooled Population
Description: as for outcome 18
Time Frame: Baseline, Week 10
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 109 | 217 | 225
Score on a scale | -1.4 (0.2) | -1.6 (0.2) | -1.9 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 1, Mixed Model for Repeated Measures — p-value has been adjusted for multiplicity; [statistical method as in outcome 16, analysis 1]; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.0 to 0.0] — Mean difference was calculated as etrolizumab arm minus placebo arm
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 17, analysis 2]; Test type: Superiority; p = 1, Mixed Model for Repeated Measures — p-value has been adjusted for multiplicity; [statistical method as in outcome 16, analysis 1]; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.7 to 0.1] — Mean difference was calculated as etrolizumab arm minus adalimumab arm

20. Secondary Outcome: Percentage of Participants in Clinical Remission at Week 10, as Determined by the MCS, GA28948 Population
Description: The Mayo Clinic Score (MCS) ranges from 0 to 12 and is a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and physician's global assessment (PGA) subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease. Clinical remission was defined as MCS less than or equal to (≤)2 with individual subscores ≤1. Participants were also classified as non-remitters if Week 10 assessments were missing or if they had received permitted/prohibited rescue therapy prior to assessment. Participants were stratified by concomitant treatment with corticosteroids or immunosuppressants at randomization and disease activity measured during screening (MCS ≤9/MCS ≥10). The Cochran-Mantel-Haenszel test adjusted the differences in remission rates and associated 95% confidence intervals for the stratification factors.
Time Frame: Week 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 72 | 142 | 144
Percentage of participants | 8.3 [3.88 to 17.01] | 23.9 [17.67 to 31.59] | 19.4 [13.81 to 26.67]
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0364, Cochran-Mantel-Haenszel — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = 10.9, 95% CI 2-sided [-0.08 to 19.48] — Difference in remission rates was calculated as the etrolizumab arm minus the placebo arm
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3383, Cochran-Mantel-Haenszel — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = -4.5, 95% CI 2-sided [-14.10 to 5.07] — Difference in remission rates was calculated as the etrolizumab arm minus the adalimumab arm

21. Secondary Outcome: Percentage of Participants in Remission at Week 10 and Week 14, as Determined by the MCS, GA28948 Population
Description: The Mayo Clinic Score (MCS) ranges from 0 to 12 and is a composite of the four following assessments of disease activity: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, and physician's global assessment (PGA) subscore. Each of the four assessments was rated with a score from 0 to 3, with higher scores indicating more severe disease. Remission was defined as MCS less than or equal to (≤)2 with individual subscores ≤1 and a rectal bleeding subscore of 0. Participants were also classified as non-remitters if Week 10 or 14 assessments were missing or the participant received permitted/prohibited rescue therapy prior to assessment. Participants were stratified by concomitant treatment with corticosteroids or immunosuppressants at randomization and disease activity measured during screening (MCS ≤9/MCS ≥10). The Cochran-Mantel-Haenszel test adjusted the differences in remission rates and associated 95% confidence intervals for the stratification factors.
Time Frame: Weeks 10 and 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 72 | 142 | 144
Percentage of participants | 2.8 [0.77 to 9.57] | 12.7 [8.17 to 19.15] | 9.0 [5.35 to 14.83]
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0900, Cochran-Mantel-Haenszel — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = 6.2, 95% CI 2-sided [-3.33 to 12.30] — Difference in remission rates was calculated as the etrolizumab arm minus the placebo arm
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3217, Cochran-Mantel-Haenszel — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 1, analysis 1]; Difference in Remission Rates = -3.6, 95% CI 2-sided [-11.07 to 3.78] — Difference in remission rates was calculated as the etrolizumab arm minus the adalimumab arm

22. Secondary Outcome: Change From Baseline in Health-Related Quality of Life at Week 10, as Assessed by the Total Inflammatory Bowel Disease Questionnaire (IBDQ) Score, GA28948 Population
Description: The IBDQ is a 32-item questionnaire containing four domains: bowel symptoms (10 items), systemic symptoms (5 items), emotional function (12 items), and social function (5 items). An overall total IBDQ score was computed by summing the individual 32-item scores. The range for the IBDQ total score is 32 to 224, with higher scores denoting better health-related quality of life. The unadjusted mean and standard deviation for each study arm are reported. The change from baseline in the IBDQ score was analyzed using an ANCOVA model taking the stratification factors used at randomization into account (concomitant treatment with corticosteroids or immunosuppressants at randomization and disease activity measured during screening [MCS ≤9/MCS ≥10]), and the baseline IBDQ score used as a covariate.
Time Frame: Baseline, Week 10
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 63 | 127 | 124
Score on a scale | 38.4 (35.7) | 39.2 (32.8) | 39.8 (35.3)
Statistical Analysis 1: Comparison: Placebo vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7919, ANCOVA — Nominal p-value; it has not been adjusted for multiplicity; Model adjusted for concomitant treatment with corticosteroids or immunosuppressants at baseline (BL), MCS (≤9 or ≥10) at BL, and IBDQ score at BL; Difference in Adjusted Means = 1.3, 95% CI 2-sided [-8.3 to 10.8] — Mean difference was calculated as etrolizumab arm minus placebo arm
Statistical Analysis 2: Comparison: Adalimumab vs Etrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8327, ANCOVA — Nominal p-value; it has not been adjusted for multiplicity; [statistical method as in outcome 22, analysis 1]; Difference in Adjusted Means = -0.8, 95% CI 2-sided [-8.7 to 7.0] — Mean difference was calculated as etrolizumab arm minus adalimumab arm

23. Secondary Outcome: Pharmacokinetics of Etrolizumab: Serum Concentration, GA28948 Population
Description: Serum concentrations of etrolizumab were evaluated at the primary endpoint visit (Week 10) and the secondary endpoint visit (Week 14). Both time points were two weeks after the most recent dose.
Time Frame: Weeks 10 and 14
Population: GA28948 Pharmacokinetics Evaluable Population: includes participants in study GA28948 who had received at least one dose of study drug and had at least one quantifiable concentration measured post-baseline. Only participants who were treated with etrolizumab were included in this analysis.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Arm/Group | Etrolizumab
Number analyzed (Participants) | 143
micrograms per millilitre (μg/mL)
  Week 10: number analyzed (Participants) | 142
  Week 10 | 13.0 (5.84)
  Week 14: number analyzed (Participants) | 12
  Week 14 | 17.1 (8.10)

24. Secondary Outcome: Number and Percentage of Participants With at Least One Adverse Event by Severity, According to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI CTCAE v4.0), GA28948 Population
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation in which a patient is administered a pharmaceutical product, regardless of causal attribution. The investigator independently assessed the severity and seriousness of each recorded AE. The AE severity grading scale for the NCI CTCAE v4.0 was used for assessing severity; any AE not specifically listed was rated according to the following grading scale from 1 to 5: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death. AEs of special interest included: elevated AST/ALT in combination with either elevated bilirubin or clinical jaundice; suspected transmission of infectious agent by the study drug; anaphylactic, anaphylactoid and systemic hypersensitivity reactions; and neurological signs, symptoms, and AEs that may suggest possible progressive multifocal leukoencephalopathy (PML).
Time Frame: From Baseline until the end of study (up to 26 weeks)
Population: GA28948 Safety Population: includes all participants in study GA28948 who received at least one dose of study drug, with participants grouped according to the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 72 | 142 | 144
Participants
  Any Adverse Event (AE) | 26 | 61 | 50
  AE with Fatal Outcome | 0 | 0 | 1
  Serious AE | 2 | 3 | 8
  AE Leading to Study Treatment Discontinuation | 0 | 2 | 2
  AE Leading to Dose Interruption | 0 | 1 | 3
  Related AE | 4 | 14 | 10
  AE by Worst Severity, Grade 1 | 11 | 33 | 21
  AE by Worst Severity, Grade 2 | 13 | 22 | 18
  AE by Worst Severity, Grade 3 | 2 | 6 | 9
  AE by Worst Severity, Grade 4 | 0 | 0 | 1
  AE by Worst Severity, Grade 5 | 0 | 0 | 1
  Any AEs of Special Interest | 0 | 0 | 0
  Confirmed PML | 0 | 0 | 0
  Infections | 7 | 17 | 15
  Serious Infections | 2 | 0 | 2
  Gastrointestinal Infections | 1 | 0 | 1
  Opportunistic Infections | 0 | 0 | 0
  Malignancies | 0 | 0 | 0
  Injection Site Reactions | 0 | 4 | 1

25. Secondary Outcome: Number and Percentage of Participants by Marked Laboratory Abnormality Status for Hematology Parameters as a Shift Table From Baseline to Week 10, GA28948 Population
Description: Laboratory tests for hematology parameters were performed and values were compared with the Roche marked reference range. A marked abnormality was defined as a test result that was outside of the Roche marked reference range (labelled as 'High' or 'Low') and represented a clinically significant change from baseline. Not every laboratory abnormality qualified as an adverse event. A laboratory test result must have been reported as an adverse event if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment or a medical intervention; or was clinically significant in the investigator's judgment. The results are presented as a shift from the baseline status to the Week 10 status. Baseline was defined as the last available assessment prior to first receipt of study drug. The 'missing' status only included participants with missing post-baseline values given they had a result at baseline. Abs = absolute count; Ery. = erythrocyte
Time Frame: From Baseline up to Week 10
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 72 | 142 | 144
Participants
  Eosinophils Absolute Count (Abs) - Normal to Normal | 66 | 130 | 130
  Eosinophils Abs - Normal to High | 0 | 0 | 1
  Eosinophils Abs - Normal to Missing | 6 | 11 | 9
  Eosinophils Abs - High to Normal | 0 | 1 | 4
  Hematocrit - Low to Low | 0 | 0 | 2
  Hematocrit - Low to Normal | 0 | 5 | 3
  Hematocrit - Normal to Low | 3 | 1 | 2
  Hematocrit - Normal to Normal | 63 | 122 | 124
  Hematocrit - Normal to High | 0 | 1 | 0
  Hematocrit - Normal to Missing | 6 | 13 | 12
  Hematocrit - High to Normal | 0 | 0 | 1
  Hemoglobin - Low to Low | 4 | 15 | 11
  Hemoglobin - Low to Normal | 4 | 5 | 9
  Hemoglobin - Low to Missing | 2 | 0 | 1
  Hemoglobin - Normal to Low | 6 | 2 | 5
  Hemoglobin - Normal to Normal | 52 | 109 | 110
  Hemoglobin - Normal to Missing | 4 | 11 | 8
  Lymphocytes Abs - Low to Low | 0 | 0 | 2
  Lymphocytes Abs - Low to Normal | 1 | 3 | 7
  Lymphocytes Abs - Normal to Low | 1 | 2 | 1
  Lymphocytes Abs - Normal to Normal | 64 | 126 | 125
  Lymphocytes Abs - Normal to Missing | 6 | 11 | 9
  Ery. Mean Corpuscular Volume - Normal to Normal | 66 | 129 | 132
  Ery. Mean Corpuscular Volume - Normal to Missing | 6 | 13 | 12
  Neutrophils, Total, Abs - Low to Normal | 3 | 1 | 2
  Neutrophils, Total, Abs - Normal to Low | 1 | 5 | 0
  Neutrophils, Total, Abs - Normal to Normal | 58 | 115 | 118
  Neutrophils, Total, Abs - Normal to High | 1 | 3 | 5
  Neutrophils, Total, Abs - Normal to Missing | 6 | 11 | 8
  Neutrophils, Total, Abs - High to Normal | 2 | 4 | 9
  Neutrophils, Total, Abs - High to High | 1 | 3 | 1
  Neutrophils, Total, Abs - High to Missing | 0 | 0 | 1
  Platelets - Normal to Normal | 60 | 120 | 122
  Platelets - Normal to High | 3 | 5 | 4
  Platelets - Normal to Missing | 8 | 13 | 12
  Platelets - High to Normal | 1 | 0 | 4
  Platelets - High to High | 0 | 4 | 1
  White Blood Cell Count - Low to Normal | 0 | 0 | 1
  White Blood Cell Count - Normal to Low | 1 | 3 | 2
  White Blood Cell Count - Normal to Normal | 65 | 127 | 132
  White Blood Cell Count - Normal to Missing | 6 | 11 | 9
  White Blood Cell Count - High to Normal | 0 | 1 | 0

26. Secondary Outcome: Number and Percentage of Participants by Marked Laboratory Abnormality Status for Chemistry Parameters as a Shift Table From Baseline to Week 10, GA28948 Population
Description: Laboratory tests for chemistry parameters were performed and values were compared with the Roche marked reference range. A marked abnormality was defined as a test result that was outside of the Roche marked reference range (labelled as 'High' or 'Low') and represented a clinically significant change from baseline. Not every laboratory abnormality qualified as an adverse event. A laboratory test result must have been reported as an adverse event if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment or a medical intervention; or was clinically significant in the investigator's judgment. The results are presented as a shift from the baseline status to the Week 10 status. Baseline was defined as the last available assessment prior to first receipt of study drug. The 'missing' status only included participants with missing post-baseline values given they had a result at baseline.
Time Frame: From Baseline up to Week 10
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Adalimumab | Etrolizumab
Number analyzed (Participants) | 72 | 142 | 144
Participants
  Albumin - Low to Low | 0 | 3 | 0
  Albumin - Low to Normal | 0 | 2 | 1
  Albumin - Normal to Low | 0 | 1 | 0
  Albumin - Normal to Normal | 69 | 132 | 137
  Albumin - Normal to Missing | 3 | 4 | 6
  Alkaline Phosphatase - Normal to Normal | 67 | 139 | 138
  Alkaline Phosphatase - Normal to High | 1 | 0 | 0
  Alkaline Phosphatase - Normal to Missing | 3 | 3 | 6
  Alkaline Phosphatase - High to High | 1 | 0 | 0
  Alanine Aminotransferase - Normal to Normal | 68 | 137 | 138
  Alanine Aminotransferase - Normal to High | 1 | 0 | 0
  Alanine Aminotransferase - Normal to Missing | 3 | 4 | 6
  Alanine Aminotransferase - High to Normal | 0 | 1 | 0
  Aspartate Aminotransferase - Normal to Normal | 67 | 137 | 137
  Aspartate Aminotransferase - Normal to High | 1 | 0 | 0
  Aspartate Aminotransferase - Normal to Missing | 4 | 4 | 7
  Aspartate Aminotransferase - High to Normal | 0 | 1 | 0
  Bicarbonate (CO2) - Low to Low | 0 | 0 | 1
  Bicarbonate (CO2) - Low to Normal | 1 | 3 | 1
  Bicarbonate (CO2) - Normal to Low | 8 | 9 | 6
  Bicarbonate (CO2) - Normal to Normal | 55 | 118 | 123
  Bicarbonate (CO2) - Normal to High | 0 | 0 | 1
  Bicarbonate (CO2) - Normal to Missing | 4 | 5 | 6
  Bicarbonate (CO2) - High to Normal | 4 | 5 | 6
  Bicarbonate (CO2) - High to High | 0 | 1 | 0
  Bicarbonate (CO2) - High to Missing | 0 | 1 | 0
  Blood Urea Nitrogen - Normal to Normal | 69 | 138 | 138
  Blood Urea Nitrogen - Normal to Missing | 3 | 3 | 6
  Blood Urea Nitrogen - High to Normal | 0 | 1 | 0
  Calcium - Low to Normal | 0 | 0 | 1
  Calcium - Normal to Normal | 69 | 139 | 137
  Calcium - Normal to Missing | 3 | 3 | 6
  Chloride - Low to Low | 0 | 1 | 0
  Chloride - Low to Missing | 1 | 0 | 0
  Chloride - Normal to Low | 2 | 0 | 1
  Chloride - Normal to Normal | 67 | 137 | 137
  Chloride - Normal to Missing | 2 | 4 | 6
  Creatinine - Normal to Normal | 69 | 139 | 138
  Creatinine - Normal to Missing | 3 | 3 | 6
  Direct Bilirubin - Normal to Normal | 68 | 134 | 134
  Direct Bilirubin - Normal to Missing | 4 | 8 | 10
  Potassium - Normal to Normal | 69 | 139 | 137
  Potassium - Normal to Missing | 3 | 3 | 7
  Sodium - Normal to Normal | 68 | 139 | 137
  Sodium - Normal to High | 1 | 0 | 1
  Sodium - Normal to Missing | 2 | 3 | 6
  Sodium - High to Missing | 1 | 0 | 0
  Total Bilirubin - Normal to Normal | 68 | 136 | 137
  Total Bilirubin - Normal to High | 1 | 2 | 1
  Total Bilirubin - Normal to Missing | 3 | 4 | 6
  Protein, Total - Low to Normal | 0 | 1 | 1
  Protein, Total - Normal to Low | 0 | 1 | 0
  Protein, Total - Normal to Normal | 67 | 132 | 136
  Protein, Total - Normal to High | 2 | 5 | 0
  Protein, Total - Normal to Missing | 3 | 3 | 6
  Protein, Total - High to High | 0 | 0 | 1

27. Secondary Outcome: Number and Percentage of Participants With Anti-Drug Antibodies (ADAs) to Etrolizumab at Baseline and Anytime Post-Baseline, GA28948 Population
Description: Anti-drug antibody (ADA) serum samples were collected from participants and analyzed using validated assays. Participants were considered to be ADA positive post-baseline if they were ADA negative or had missing data at baseline, but developed an ADA response following etrolizumab drug exposure (treatment-induced ADA response), or if they were ADA positive at baseline and the titer of one or more post-baseline samples was at least 0.60 titer units greater than the titer of the baseline sample (treatment-enhanced ADA response). Participants were considered to be ADA negative if they were ADA negative or had missing data at baseline and all post-baseline samples were negative, or if they were ADA positive at baseline but did not have any post-baseline samples with a titer that was at least 0.60 titer unit greater than the titer of the baseline sample (treatment unaffected).
Time Frame: Pre-dose (0 hour) on Day 1 and Week 4, Week 10, Week 14, and early termination/end of safety follow-up (up to 26 weeks)
Population: GA28948 Safety Population: includes all participants in study GA28948 who received at least one dose of study drug, with participants grouped according to the treatment received. The analysis of ADAs at baseline and post-baseline only included participants who received treatment with etrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Etrolizumab
Number analyzed (Participants) | 144
Participants
  Positive for ADAs at Baseline (BL) | 6
  Negative for ADAs at BL | 138
  Post-BL: Positive for Treatment Emergent ADAs | 27
  Post-BL ADA Positive: Treatment-Induced ADAs | 27
  Post-BL ADA Positive: Treatment-Enhanced ADAs | 0
  Post-BL: Negative for Treatment Emergent ADAs | 117
  Post-BL ADA Negative: Treatment Unaffected | 6

ADVERSE EVENTS:
Time Frame: From Baseline until the end of study (up to 26 weeks)
Description: The adverse events reported here are those that occurred only in participants enrolled in study GA28948 who received at least one dose of study drug. For the adverse events that occurred in participants enrolled in the identically designed study, GA28949, please refer to its study record, NCT02171429.
Arm/Group | Placebo | Adalimumab | Etrolizumab
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/142 | 1/144
Serious Adverse Events (participants affected / at risk) | 2/72 | 3/142 | 8/144
Other Adverse Events (participants affected / at risk) | 7/72 | 17/142 | 6/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=72) | Adalimumab (N=142) | Etrolizumab (N=144)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Eye infection toxoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=72) | Adalimumab (N=142) | Etrolizumab (N=144)
Colitis ulcerative (Gastrointestinal disorders) | 4 (4) | 8 (9) | 5 (5)
Headache (Nervous system disorders) | 3 (4) | 9 (15) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT02163759/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT02163759/SAP_001.pdf